CLINICAL TRIAL: NCT03934398
Title: Be-HealthY: Behavioral Risk Factors for Poor Vascular Health in Youth
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00196923; 1R56HL139620 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Prehypertension; Hypertension; Overweight and Obesity; Elevated Blood Pressure; Endothelial Dysfunction; Vascular Stiffness; Sleep
MeSH Terms: conditions — Prehypertension; Hypertension; Overweight; Obesity | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ReNEW Clinical Cohort: Individuals evaluated in the ReNEW Clinic at Johns Hopkins University who join the ReNEW Clinic Cohort Study are eligible for this cross-sectional study. Tests will be done for all participants which includes Cardiovascular Assessments, Actigraphy and Laboratory assessments.
  Interventions: Diagnostic Test: Cardiovascular Assessments; Diagnostic Test: Actigraphy; Diagnostic Test: Laboratory assessments; Diagnostic Test: Emotional/Behavioral Assessments

INTERVENTIONS:
Diagnostic Test: Cardiovascular Assessments — Participants will undergo the following cardiovascular assessments: 24-hour blood pressure monitoring, arterial stiffness measurements, endothelial function measurements.
Diagnostic Test: Actigraphy — Participants will wear an actigraph device for 7 days to measure participant's activity and sleep.
Diagnostic Test: Laboratory assessments — Participants will provide blood and urine samples for laboratory assessments.
Diagnostic Test: Emotional/Behavioral Assessments — Participants and parents will fill out questionnaires for emotional/behavioral assessments

SUMMARY:
The investigators aim to determine the association of dietary intake on cardiovascular disease risk factors among children with overweight and obesity who are being evaluated for elevated blood pressure.

The investigators will also investigate for predictors of vascular function and determine if predictors vary by level of sodium intake.

DETAILED DESCRIPTION:
This research is being done to determine if the food or salt eaten can cause arteries to be stiffer and/or not work as well and if it can impact blood pressure over a 24-hour period of time. The investigators also want to determine if there are any risk factors or blood tests that can predict how stiff arteries are or how well arteries function. The investigators hope that the information from this study will help the investigators prevent blood pressure-related cardiovascular disease in children. This knowledge could help shape future guidelines on how to best prevent and treat high blood pressure and heart disease in children.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Elevated blood pressure
* Referred to the ReNEW Clinic at Johns Hopkins University for evaluation and treatment of elevated blood pressure.

Exclusion Criteria:

* The only children who will not be eligible for inclusion in this study are those who are non-English speaking.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults up to 22 years of age who have overweight or obesity and elevated blood pressure, and were referred to the ReNEW Clinic for evaluation and treatment of elevated blood pressure.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness as assessed by Pulse wave velocity | 1 day
  This will be determined from Pulse wave velocity (m/sec) done at the study visit
Arterial stiffness as assessed by Ambulatory Arterial Stiffness Index (AASI) | 1 day
  The Ambulatory Arterial Stiffness Index will be determined from data obtained from vascular measures and during 24-hour ambulatory blood pressure monitoring. Arterial stiffness increases as the regression slope approaches 0 and the AASI approaches 1.
Arterial stiffness as assessed by Augmentation Index | 1 day
  The Augmentation Index (measured as a percentage) will be determined from a vascular assessment and data obtained during 24-hour ambulatory blood pressure monitoring. A greater Augmentation Index represents a stiffer, less compliant vessel.
Endothelial function as assessed by Laser Doppler flow perfusion | 1 day
  The percent change in mean blood flow will be determined from Laser Doppler flow perfusion measurements obtained using a heating protocol.
Mean Blood pressure (mmHg) | 1 day
  Mean daytime systolic blood pressure in millimeters of mercury (mmHg) will be determined from 24-hour blood pressure monitoring.

SECONDARY OUTCOMES:
Pediatric Adverse Childhood Events (ACEs) score | 1 day
  The Pediatric ACEs questionnaire contains 17 yes or no questions about stressful or traumatic life events. Greater exposure to adverse childhood experiences (ACEs) is associated with poorer physical and mental health. Some researchers have suggested that an ACEs score of greater than or equal to 3 or 4 significantly increases the risk for health problems, however, there is no widely accepted threshold for how many ACEs endorsed is clinically significant or more predictive of these problems.
Children's Emotion Management Scale (CEMS) score | 1 day
  The Children's Emotional management scale is a questionnaire that consists of 33 questions (3 point Likert scale) examining youth's ability to regulate appropriately their negative emotions (i.e. anger, sadness, and worry). Generally, poorer emotion regulation capabilities are associated with poorer health outcomes, with most research looking at CV outcomes in adults.
Behavior Assessment for Children (BASC) score | 1 day
  The Behavior Assessment for Children is a questionnaire that consists of 189 questions (True/False and 4 point Likert scale). It is a broad behavioral screening measure commonly used in child and adolescent psychology and psychiatric settings.It has three primary scales: internalizing (e.g., depression, anxiety), externalizing (e.g., aggression, hyperactivity), and total problems (combination of internalizing and externalizing plus attention problems and withdrawal subscales). Scores between 60-69 are considered "at risk" for clinical problems and scores of 70+ are considered clinically significant presence of those symptoms. Any scores that are not in this range are considered to be within normal limits and not indicative of difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy M Brady, M.D., PhD., Principal Investigator — Johns Hopkins University Division of Pediatric Nephrology
Locations (1):
- Johns Hopkins School of Medicine Division of Pediatric Nephrology, Baltimore, Maryland, United States